CLINICAL TRIAL: NCT03146741
Title: Open-Labeled Trial Of Zepatier For Treatment Of Hepatitis C-Negative Patients Who Receive Heart Transplants From Hepatitis C-Positive Donors
Brief Title: Zepatier For Treatment Of Hepatitis C-Negative Patients Who Receive Heart Transplants From Hepatitis C-Positive Donors (HCV)
Acronym: USHER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 826708
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Results first posted 2020-02-26 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zepatier (grazoprevir 100mg and elbasvir 50 mg) (Experimental)
  Interventions: Drug: Zepatier

INTERVENTIONS:
Drug: Zepatier — Zepatier (grazoprevir 100mg and elbasvir 50 mg once daily) is taken by mouth for 12 weeks unless a genetic variation is detected. In this case treatment with Zepatier will be extended to 16 weeks. Study subjects with treatment failure will be provided open-label Zepatier + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.

SUMMARY:
This study is being conducted to determine safety and effectiveness of transplanting hearts from Hepatitis C-positive donors into Hepatitis C-negative patients on the heart transplant waitlist, who will then be treated with Zepatier after transplantation.

DETAILED DESCRIPTION:
Open-labelled pilot clinical trial of Zepatier (MK-5172 and MK-8742/Grazoprevir + Elbasvir) in at least 20 HCV-negative subjects receiving a heart transplant from a HCV-positive donor. Eligible subjects will receive a heart transplant from a deceased-donor with genotype 1 or 4 HCV, and then will receive 12 weeks of Zepatier after heart transplantation when infection with HCV is confirmed in these heart transplant recipients. Treatment will be complete after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Class III or IV CHF refractory to maximal medical therapy (ACE inhibitor, B-blocker, digoxin and diuretics, resynchronization therapy or Implantable Cardioverter Defibrillator when applicable) and/or conventional surgery.
* Inoperable coronary artery disease with intractable anginal symptoms
* Malignant ventricular arrhythmias unresponsive to medical or surgical therapy
* 18-65 years of age
* Obtained agreement for participation from the transplant cardiology team
* No evident contraindication to liver transplantation other than the underlying cardiac disorder
* Able to travel to the University of Pennsylvania for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
* No active illicit substance abuse
* Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant due to the increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method of birth control or remain abstinent following transplant due to risk of HCV transmission
* Inclusion criteria for treatment (not for entry as study patient) will include any detectable HCV RNA by week 4 post-heart transplantation
* Able to provide informed consent

Exclusion Criteria:

* Hepatocellular carcinoma
* HIV positive
* HCV antibody positive and/or RNA positive
* Hepatitis B surface antigen, core antibody, and/or DNA positive
* Any other chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD) with abnormal liver enzymes
* Persistently elevated liver transaminases
* Congenital heart disease
* Fibrosis by liver biopsy or total bilirubin > 2.5 with associated evidence of synthetic dysfunction.
* Pregnant or nursing (lactating) women
* Known allergy or intolerance to tacrolimus that would require post-transplant administration of cyclosporine, rather than tacrolimus given the drug-drug interaction between cyclosporine and ZEPATIER
* Waitlisted for a multi-organ transplant
* Evidence of end organ damage due to diabetes (e.g. retinopathy, nephropathy, ulcerations) and /or brittle diabetes mellitus (e.g. history of diabetic ketoacidosis) and/or uncontrolled diabetes as evidence by a HgbA1C of 7.5-8.5.
* Chronic bronchitis, chronic obstructive pulmonary disease, inability to stop smoking.
* Hematologic: Significant coagulation abnormalities, bleeding diatheses.
* Psychosocial: Profound neurocognitive impairment with absence of social support.
* Active mental illness or psychosocial instability
* Inadequate insurance or financial support for post-transplant care.
* Evidence of drug, tobacco or alcohol abuse within the past six months and completion of recommended therapy/services or meets satisfied parameters as indicated by social work staff and/or consult team.
* History of chronic non-compliance.
* Amyloidosis (restricted to cardiac only, without evidence of extra cardiac involvement)
* BMI ≥38
* Active peptic ulcer disease.
* Severe malnutrition.
* Major chronic disabling illness (e.g. lupus, severe arthritis, neurologic diseases, previous stroke with profound residual).
* Pulmonary infarction within the past 6 weeks
* Severe pulmonary hypertension as evidenced by a fixed pulmonary vascular resistance of greater than 4 Wood units on appropriate medical therapy.
* Patient refusal to receive blood products or transfusions during heart transplant surgery.
* Severe chronic obstructive pulmonary disease
* Current clinical sepsis.
* Symptomatic or severe vascular disease.
* Chronic Kidney Disease Stage IV, Glomerular Filtration Rate < 30
* History of Mantle radiation.
* Asymptomatic renal cell carcinoma <1 year from curative treatment.
* Symptomatic renal cell carcinoma <5 years from curative treatment.
* Prostate cancer <2 years from curative treatment.
* Uterine or cervical cancer <2 years from curative treatment.
* Any other cancer other than the above including malignant melanoma, < 5 years from treatment apart from other skin malignancies.

Donor Organ Selection Criteria:

General criteria (although there can be exceptions on a case-by-case basis)

* Detectable HCV RNA
* Genotype 1 or 4 HCV
* Age <=55 years
* No history of coronary artery disease
* No congenital heart disease except a repaired atrial septal defect (ASD) provided the patient has normal right ventricular function
* No history of arrhythmia (atrial fibrilation, atrial flutter or VT) except during resuscitation from fatal event.
* No evidence of cirrhosis

Echocardiographic criteria:

* Left ventricular ejection fraction (LVEF) >=50%
* Normal right ventricular function
* No left ventricular hypertrophy (LVH) - septal wall thickness <1 cm
* No left ventricular hypertrophy (LVH)- posterior wall thickness <1 cm
* No significant valvular heart disease - more than mild tricuspid regurgitation, more than mild mitral regurgitation, more than trace aortic regurgitation. No mitral or aortic stenosis.
* No congenital heart disease - transposition of the great vessels, ventricular septal defect (VSD), ASD, and/or single ventricle (Fontan)

Right heart catheterization criteria:

* Right atrial pressure <=10mmHg
* Pulmonary capillary wedge pressure <=18mmHg
* CI >=2.1 l/min/m2
* Pulmonary hypertension is allowed if the patient has normal right ventricular function and a normal tricuspid valve

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reese, MD, MSCE, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sulkowski M, Hezode C, Gerstoft J, Vierling JM, Mallolas J, Pol S, Kugelmas M, Murillo A, Weis N, Nahass R, Shibolet O, Serfaty L, Bourliere M, DeJesus E, Zuckerman E, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 8 weeks versus 12 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin in patients with hepatitis C virus genotype 1 mono-infection and HIV/hepatitis C virus co-infection (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1087-97. doi: 10.1016/S0140-6736(14)61793-1. Epub 2014 Nov 11. PMID 25467560
- [Background] Lawitz E, Gane E, Pearlman B, Tam E, Ghesquiere W, Guyader D, Alric L, Bronowicki JP, Lester L, Sievert W, Ghalib R, Balart L, Sund F, Lagging M, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 12 weeks versus 18 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin for hepatitis C virus genotype 1 infection in previously untreated patients with cirrhosis and patients with previous null response with or without cirrhosis (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1075-86. doi: 10.1016/S0140-6736(14)61795-5. Epub 2014 Nov 11. PMID 25467591
- [Background] Forns X, Gordon SC, Zuckerman E, Lawitz E, Calleja JL, Hofer H, Gilbert C, Palcza J, Howe AY, DiNubile MJ, Robertson MN, Wahl J, Barr E, Buti M. Grazoprevir and elbasvir plus ribavirin for chronic HCV genotype-1 infection after failure of combination therapy containing a direct-acting antiviral agent. J Hepatol. 2015 Sep;63(3):564-72. doi: 10.1016/j.jhep.2015.04.009. Epub 2015 Apr 18. PMID 25895428
- [Background] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356
- [Background] O'Leary JG, Neri MA, Trotter JF, Davis GL, Klintmalm GB. Utilization of hepatitis C antibody-positive livers: genotype dominance is virally determined. Transpl Int. 2012 Aug;25(8):825-9. doi: 10.1111/j.1432-2277.2012.01498.x. Epub 2012 May 30. PMID 22643162
- [Background] Reese PP, Abt PL, Blumberg EA, Goldberg DS. Transplanting Hepatitis C-Positive Kidneys. N Engl J Med. 2015 Jul 23;373(4):303-5. doi: 10.1056/NEJMp1505074. No abstract available. PMID 26200976
- [Background] Reddy KR FS, et al. Ledipasvir/Sofosbuvir with Ribavirin for the Treatment of HCV in Patients with Post Transplant Recurrence: Preliminary Results of a Prospective, Multicenter Study. Hepatology. 2014;60:200A.
- [Background] Roth D, Nelson DR, Bruchfeld A, Liapakis A, Silva M, Monsour H Jr, Martin P, Pol S, Londono MC, Hassanein T, Zamor PJ, Zuckerman E, Wan S, Jackson B, Nguyen BY, Robertson M, Barr E, Wahl J, Greaves W. Grazoprevir plus elbasvir in treatment-naive and treatment-experienced patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease (the C-SURFER study): a combination phase 3 study. Lancet. 2015 Oct 17;386(10003):1537-45. doi: 10.1016/S0140-6736(15)00349-9. Epub 2015 Oct 5. PMID 26456905
- [Background] Van Deerlin, V. (December 2015). Hepatitis C Virus Genotyping (GenMark Assay) Validation Summary.
- [Background] Pawlak R RJ, Maranan G, Michel-Treil V, Schutzbank T. A Comparative Evaluation of the Siemens VERSANT HCV Genotype 2.0 (LiPA) and GenMark eSensor HCV Direct Genotyping Tests. CVS 2013 Covance; 2013
- [Background] Dahl A HD, Ogorek T, Hansen G. Comparison of the GenMark Direct Genotype Assay with the LiPA Genotype Assay Using a Diverse Spectrum of HCV Clinical Samples Encountered in a High Risk Inner City HCV Population. CVS 2013 Hennepin; 2013.
- [Background] Woodberry M SK, Castor J, Cook L, Jerome K. Genotyping of Hepatitis C Virus by the Genmark DX Esensor HCVG Direct Test. CVS 2013 UW-Seattle 2013
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute. (June 2010). Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
- [Background] Merck Sharp & Dohme Corporation (January 2016). ZEPATIER™ tablets. Highlights of Prescribing Information. 2016.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Elbasvir (MK-8742). Investigator's Brochure (8th Ed.). 2015.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Grazoprevir (MK-5172). Investigator's Brochure (10th Ed.). 2015.

RESULTS

PARTICIPANT FLOW:
Groups:
- Zepatier (Grazoprevir 100mg and Elbasvir 50 mg): Zepatier (grazoprevir 100mg and elbasvir 50 mg once daily) is taken by mouth for 12 weeks unless a genetic variation is detected. In this case treatment with Zepatier will be extended to 16 weeks. Study subjects with treatment failure will be provided open-label Zepatier + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.
Period: Overall Study
Arm/Group | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg)
Started | 20
Completed | 10
Not Completed | 10
Not completed — Txp with non-HCV+ heart | 4
Not completed — Listeted for MOT | 2
Not completed — Physician Decision | 2
Not completed — Awaiting txp | 2

BASELINE CHARACTERISTICS:
Arm/Group | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg)
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.5 [45 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-treatment Sustained Virologic Response (SVR)
Description: The primary analysis will be based on a calculation of SVR rates (number of subjects with SVR; negative HCV RNA after completing Zepatier therapy) / (number of subjects treated with Zepatier post-heart transplantation)
Time Frame: Baseline to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg)
Number analyzed (Participants) | 10
Participants | 9

2. Primary Outcome: Number of Severe Adverse Events (SAE) Attributable to HCV Therapy Post-heart Transplant
Time Frame: Baseline to 52 weeks
Measure: Number; unit: Severe adverse event
Arm/Group | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg)
Number analyzed (Participants) | 10
Severe adverse event | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Zepatier (Grazoprevir 100mg and Elbasvir 50 mg): Zepatier (grazoprevir 100mg and elbasvir 50 mg once daily) is taken by mouth for 12 weeks unless a genetic variation is detected - in this case treatment with Zepatier will be extended to 16 weeks. Study subjects with treatment failure will be provided open-label Zepatier + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.
  Note: No subjects experienced treatment failure requiring sofosbuvir. Adverse events were collected the same way for all subjects in the setting of only 1 medication regimen intervention (Zepatier). For that reason we present the results and AEs in 1 arm containing all 10 subjects.
Arm/Group | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg) (N=10)
Death (Cardiac disorders) | 1
Post-op re-intubation (Surgical and medical procedures) | 2
Abdominal infection (Gastrointestinal disorders) | 1
CMV (Infections and infestations) | 1
Hemorrhagic shock (General disorders) | 1
Terminal ileun ulcer (Gastrointestinal disorders) | 1
Fall (Psychiatric disorders) | 1
Non-infective gastroenteritis and colitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zepatier (Grazoprevir 100mg and Elbasvir 50 mg) (N=10)
Headache (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03146741/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03146741/ICF_001.pdf